CLINICAL TRIAL: NCT05258994
Title: Early Care and Education Leadership Study: Descriptive Study
Acronym: ExCELS
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); University of Massachusetts, Boston (Other)
Responsible Party: Sponsor
Other Study IDs: 50708
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Leadership in Early Care and Education Centers
Keywords: Leadership; Infant-toddler care; Early child development; Early childhood education; Head Start; Child care; Day care; Preschool; Child care and early education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mathematica and the Institute for Early Education Leadership and Innovation at the University of Massachusetts Boston, conducted a descriptive study within the Early Care and Education Leadership Study (ExCELS). ExCELS is funded by the Office of Planning, Research, and Evaluation within the Administration for Children and Families in the U.S. Department of Health and Human Services. The goal of the descriptive study is to develop a new measure of early care and education (ECE) leadership that has strong psychometric properties and examines associations among key constructs and outcomes on how ECE leadership could support quality improvements. In early 2022, the study team recruited 132 ECE centers serving children whose ages range from birth to age 5 (but who are not yet in kindergarten) and supported by Head Start grants or Child Care Development Fund subsidies. In spring 2022, the study team conducted phone interviews to collect center characteristics and learn about the center's staffing structure and leadership positions, and distributed surveys to center managers and teaching staff in recruited centers.

DETAILED DESCRIPTION:
Leadership is widely recognized as an essential driver of organizational performance and improvement, but little is known about its role in driving the quality of care and education centers provide and outcomes for staff, children, and families. ExCELS seeks to fill the definitional and measurement gaps to help the early childhood field understand how effective leaders can improve quality experiences for children in early care and education (ECE) settings.

The ExCELS descriptive study includes a purposive sample of 132 ECE centers from four states. These selected four states vary on administrator qualifications; quality rating and improvement system (QRIS) participation levels; licensing requirements to reflect the regulatory environment; funding sources (e.g., Child Care and Development Fund (CCDF) or Head Start funding) to support access and quality; and geographic diversity. Within each selected state, centers were selected to achieve variability in funding sources, center size, and geography. The study includes ECE centers serving children whose ages range from birth to age 5 (but who are not yet in kindergarten) who receive at least 20 percent of their funding from Head Start grants or CCDF subsidies.

The study team conducted the following activities with the recruited centers:

1. An engagement interview with the primary site leader (the person in the building who is responsible for oversight of all that happens in the center on a daily basis) to collect center characteristics and confirm center eligibility for the study
2. A staffing structure and leadership positions interview with the primary site leader to understand the staffing structure and formal leadership positions at the center, and
3. Surveys of center managers and teaching staff to understand key leadership elements related to the care and education of young children (on who participates in decision-making, their values and beliefs, and what they do to support high quality practices, coordination among staff and with families, having a shared vision, along with efficient operations), the center's culture, climate, and communication (such as collaboration among staff or whether there is a culture of respect, shared growth, and learning), and outcomes for the center and staff (job satisfaction, staff well-being and mental health, and staff retention).

ELIGIBILITY:
Inclusion Criteria:

* Early care and education (ECE) centers serving children whose ages range from birth to age 5, not yet in kindergarten, who are supported by Head Start or Child Care and Development Fund (CCDF) subsidies. A center is defined as a specific physical location where ECE is delivered to children whose ages range from birth to age 5 (not yet in kindergarten) with at least two classrooms.

Exclusion Criteria:

* Classrooms operated by public schools
* Centers offering less than four hours of early childcare education each day
* Drop-in child care settings

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Center-based early care and education settings that receive at least 20 percent of its funding from Head Start or the Child Care and Development Fund (CCDF) and serve children whose ages range from birth to age 5 (not yet in kindergarten). Data collection included interviews with each center's primary site leader (the person in the building who is responsible for oversight of all that happens in the center on a daily basis) and surveys for select center managers and all teaching staff.
Sampling Method: Non-Probability Sample
Enrollment: 1164 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Job Satisfaction | 5 months
  Study-developed survey on job commitment (intention to continue to work at center); and satisfaction (enjoy job, make a difference, choose career again)
Staff well-being and mental health | 5 months
  Job stress; four-item scale with response options from strongly disagree to strongly agree with the stronger agreement indicating more job stress (Institute of Behavioral Research. (2005). TCU Survey of Organizational Functioning (TCU SOF). Fort Worth: Texas Christian University, Institute of Behavioral Research. Available at ibr.tcu.edu.)
Staff retention | 5 months
  Study-developed survey on teaching staff turnover over past 12 months
Teaching staff report of family involvement | 5 months
  Parent involvement measure from Essential 0-5 Survey (Ehrlich, Stacy B., Debra M. Pacchiano, Amanda G. Stein, Maureen R. Wagner, Stuart Luppescu, Sangyoon Park, Elizabeth Frank, Holly Lewandowski, and Christopher Young. "Organizing Early Education for Improvement: Testing a New Survey Tool." Chicago, IL: University of Chicago Consortium on School Research and the Ounce of Prevention Fund, 2018.)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Kirby, M.P.P., Study Director — Mathematica Policy Research, Inc.; Lizabeth Malone, Ph.D., Principal Investigator — Mathematica Policy Research, Inc.; Anne Douglass, Ph.D., Principal Investigator — University of Massachusetts, Boston
Locations (1):
- Mathematica, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team plans to archive a restricted-use data file at the Child and Family Data Archive for secondary analysis by qualified researchers. The study team will implement procedures to ensure that data are prepared in accordance with archive requirements, removing all linkable identifiers and geographic details as well as all open-ended text and verbatim responses from all data files.
Time Frame: Data will become available within 1 year of completion.
Access Criteria: Applications for access to restricted-use data file include completing and adhering to a User Agreement.
URL: https://doi.org/10.3886/ICPSR38706

REFERENCES:
- [Background] G. Kirby, A. Douglass, J. Lyskawa, C. Jones, and L. Malone. (2021). Understanding Leadership in Early Care and Education: A literature review. OPRE Report 2021-02. Washington, DC: Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- See also: Early Care and Education Leadership Study (ExCELS), 2018-2023 - Overview — https://www.acf.hhs.gov/opre/project/early-care-and-education-leadership-study-excels-2018-2023
- See also: Mathematica: Early Care and Education Leadership Study (ExCELS) 2018-2023 — https://mathematica.org/projects/early-care-and-education-leadership-study-excels